CLINICAL TRIAL: NCT04706169
Title: Age-related Differences in Motor Recruitment Patterns of the Shoulder in Dynamic and Isometric Contractions. A Cross-sectional Study
Brief Title: Age-related Differences in Shoulder Dynamic and Isometric Contractions
Status: Completed | Type: Observational
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: University of Alcala (Other)
Responsible Party: Principal Investigator, Cristina Lirio, Principal Investigator, PhD, University of Castilla-La Mancha
Other Study IDs: CLirio04
Record Dates: First submitted 2021-01-09; First posted 2021-01-12 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Electromyography
Keywords: Age groups; Shoulder muscles; Musculoskeletal diseases
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Electromyography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Older adults: Participants, without symptoms in the shoulder and / or cervical area (at least the last year), were assigned to the Older adult group: over 65 years.
  Interventions: Device: Surface Electromyography
- Adults: Participants, without symptoms in the shoulder and / or cervical area (at least the last year), were assigned to the Adult groups: 20 to 64 years.
  Interventions: Device: Surface Electromyography

INTERVENTIONS:
Device: Surface Electromyography — SEMG was used to measure the amplitude and onset of five shoulder muscle electrical signal, performing glenohumeral abduction. In this movement, the middle deltoid muscle was selected because it is a main motor. The infraspinatus muscle represented the rotator cuff muscle group. The middle deltoid muscle was selected as the representative of shoulder abduction because it is a main motor in this movement. The trapezius muscle and the serratus anterior muscle were chosen as representative established of the ascending scapular rotator muscles.

SUMMARY:
A cross-sectional descriptive study, in which the surface electromyographic activity of five shoulder muscles was compared in two populations: older adults and adults. The evaluation of the electromyographic data offers a suitable foundation to understand aging process.

This supports that surface electromyography provide information about the aged shoulder muscles. Loss of functionality is suffered by a high percentage of older adults, which greatly limits their physical activity. In this sense, this paper presents findings that might be related with possible therapeutic approaches in subsequent studies.

DETAILED DESCRIPTION:
Aging processes in the musculoskeletal system lead to functional impairments that restrict participation. Purpose: To assess differences in force and motor recruitment patterns of shoulder muscles between age groups to understand functional disorders. A cross-sectional study comparing thirty adults (20-64) and 30 older adults (>65). Surface-electromyography (sEMG) of the middle deltoid, upper and lower trapezius, infraspinatus and serratus anterior muscles was recorded. Maximum isometric voluntary contraction (MIVC) was determined at 45° glenohumeral abduction. For the sEMG signal registration, concentric and excentric contraction with and without 1 kg and isometric contraction were requested. Participants abducted the arm from 0° up to an abduction angle of 135° for concentric and excentric contraction; and from 0º to 45º and remained there at 80% of the MIVC level while isometrically pushing against a handheld dynamometer. Differences in sEMG amplitudes (root mean square, RMS) of all contractions, but also onset latencies during concentric contraction of each muscle between age groups were analyzed. Statistical differences in strength (Adults>Older adults;0.05) existed between groups. No significant differences in RMS values of dynamic contractions were detected, except for serratus anterior, but there were for isometric contraction of all muscles analyzed (Adults>Older adults;0.05). The recruitment order varied between age groups, showing a general tendency towards delayed onset times in Older Adults, except for the upper trapezius muscle. Age differences in muscle recruitment patterns were found, which underscores the importance of developing musculoskeletal data to prevent and guide geriatric shoulder pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* No previously manifested symptoms in the shoulder joint and/or the neck during the past year,

Exclusion Criteria:

* Moderate or severe cognitive impairment
* Rheumatologic diseases
* Massive osteoarthritis
* Tumors
* Shoulder joint instability
* Circulatory disorders (hemophilia clotting problems)
* Dermatological problems exacerbated by contact with skin.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants came from Madrid and Castilla La Mancha (Spain) and voluntarily attended the Unit of the Research Group "Physical Therapy in Women´s Health Processes" in the Department of Physical Therapy, University of Alcalá, and the Ocaña Senior Center.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-12; Primary Completion 2019-01 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
The mean Root Mean Square (RMS) value | day 1
  The electromyographic data were captured simultaneously on a computer by using the LabChart® software. Within the time interval from 2 to 4 seconds after contraction initiation a power spectrum analysis was performed together with the determination of RMS values. The mean RMS values were automatically obtained from the software.
onset muscle contraction | day 1
  The onset was obtained as the time distance of the interception between the level of pre-activation relative to the onset of arm displacement during dynamic contraction and the linearly interpolated RMS slope

SECONDARY OUTCOMES:
Maximal isometric voluntary contraction | day 1
  Using hand-held dynamometer
body mass index | day 1
  is a measure of body fat based on height and weight that applies to adult men and women. Enter your weight and height using standard or metric measures.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Lirio-Romero, PhD, Principal Investigator — University of Castilla-La Mancha

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lirio-Romero C, Anders C, De La Villa-Polo P, Torres-Lacomba M. Implications on older women of age- and sex-related differences in activation patterns of shoulder muscles: A cross-sectional study. J Women Aging. 2019 Nov-Dec;31(6):492-512. doi: 10.1080/08952841.2018.1521654. Epub 2018 Sep 25. PMID 30252611
- [Background] McManus L, De Vito G, Lowery MM. Analysis and Biophysics of Surface EMG for Physiotherapists and Kinesiologists: Toward a Common Language With Rehabilitation Engineers. Front Neurol. 2020 Oct 15;11:576729. doi: 10.3389/fneur.2020.576729. eCollection 2020. PMID 33178118
- [Background] Medved V, Medved S, Kovac I. Critical Appraisal of Surface Electromyography (sEMG) as a Taught Subject and Clinical Tool in Medicine and Kinesiology. Front Neurol. 2020 Oct 26;11:560363. doi: 10.3389/fneur.2020.560363. eCollection 2020. PMID 33192993